CLINICAL TRIAL: NCT03237481
Title: A Phase 3, Randomized, Double Blind, Saline Placebo and Active Controlled, Multicenter Study of HTX 011 Via Local Administration for Postoperative Analgesia and Decreased Opioid Use Following Unilateral Open Inguinal Herniorrhaphy
Brief Title: Phase 3 Herniorrhaphy Study for Postoperative Analgesia (EPOCH 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HTX-011-302
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
Keywords: inguinal hernia; hernia; hernia surgery; postoperative pain; herniorrhaphy
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal; Hernia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Treatment Group 1: HTX-011 (Experimental): HTX 011 (bupivacaine/meloxicam)
  Interventions: Drug: HTX-011; Device: Luer-lock applicator; Device: Vial access device
- Treatment Group 2: Bupivacaine HCI (Active Comparator): Bupivacaine HCl
  Interventions: Drug: Bupivacaine HCl
- Treatment Group 3: Saline Placebo (Placebo Comparator): Saline placebo
  Interventions: Drug: Saline placebo; Device: Luer-lock applicator

INTERVENTIONS:
Drug: HTX-011 — HTX 011 (bupivacaine/meloxicam), 300 mg/9 mg by instillation
  Arms: Treatment Group 1: HTX-011
Drug: Bupivacaine HCl — Bupivacaine HCl without epinephrine, 75 mg by injection
  Arms: Treatment Group 2: Bupivacaine HCI
Drug: Saline placebo — Saline placebo by instillation
  Arms: Treatment Group 3: Saline Placebo
Device: Luer-lock applicator — Applicator for instillation
  Arms: Treatment Group 1: HTX-011; Treatment Group 3: Saline Placebo
Device: Vial access device — Device for withdrawal of drug product
  Arms: Treatment Group 1: HTX-011

SUMMARY:
This is a Phase 3, randomized, double-blind, saline placebo- and active-controlled, multicenter study to evaluate the analgesic efficacy and safety of HTX 011 administered via local administration into the surgical site in subjects undergoing unilateral open inguinal herniorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo a unilateral open inguinal herniorrhaphy with mesh under general anesthesia.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Had any prior inguinal hernia repair.
* Has a planned concurrent surgical procedure.
* Has other pre existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken NSAIDs within 10 days prior to the scheduled surgery.
* Has taken opioids within 24 hours prior to the scheduled surgery (3 days for long-acting).
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has initiated treatment with medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* Has a known history of Hepatitis B, human immunodeficiency virus (HIV), or active Hepatitis C.
* Has uncontrolled anxiety, psychiatric, or neurological disorder that, in the opinion of the Investigator, might interfere with study assessments.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention deficit/hyperactivity disorder) may be eligible for participation in the study. Subjects taking medical marijuana are not allowed to participate in the study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half lives.
* Has undergone 3 or more surgeries within 12 months.
* Has a body mass index (BMI) >39 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (22):
  - Eliza Coffee Memorial Hospital, Florence, Alabama
  - Shoals Medical Trials, Inc., Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Trovare Clinical Research, Inc., Bakersfield, California
  - Alliance Research Centers, Laguna Hills, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - HD Research Corp, Riverside, California
  - American Institute of Research, Whittier, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Cornerstone Research Institute, LLC, Longwood, Florida
  - Park Place Surgery Center, Maitland, Florida
  - University of Miami, Miami, Florida
  - St. Louis Clinical Trials, St Louis, Missouri
  - eStudySite, Las Vegas, Nevada
  - Midwest Clinical Research, Dayton, Ohio
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Westside Surgical Hospital, Houston, Texas
  - Plano Surgical Hospital, Plano, Texas
  - Endeavor Clinical Trials, P.A., San Antonio, Texas
  - EPIC Medical Research, LLC, Murray, Utah
  - Jean Brown Research, Salt Lake City, Utah
- Belgium (2):
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Ziekenhuis Oost Limburg, Genk

REFERENCES:
- [Derived] Minkowitz H, Soto R, Fanikos J, Hammer GB, Mehta N, Hu J, Redan J. Opioid-Free Recovery After Hernia Repair with HTX-011 as the Foundation of a Non-Opioid, Multimodal Analgesia Regimen in a Real-World Setting: A Randomized, Open-Label Study. Pain Ther. 2021 Dec;10(2):1295-1308. doi: 10.1007/s40122-021-00289-2. Epub 2021 Jul 27. PMID 34318438
- [Derived] Yip T, Hu J, Hawn PS, Yamamoto A, Oderda G. HTX-011 effectively reduces postoperative pain intensity and opioid use in the elderly. Pain Manag. 2022 Jan;12(1):45-57. doi: 10.2217/pmt-2021-0043. Epub 2021 Jul 21. PMID 34284613

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group 1: HTX-011: HTX-011 (bupivacaine/meloxicam), 300 mg/9 mg by instillation.
- Treatment Group 2: Bupivacaine HCI: Bupivacaine HCl without epinephrine, 75 mg by injection.
- Treatment Group 3: Saline Placebo: Saline Placebo by instillation.
Period: Overall Study
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Bupivacaine HCI | Treatment Group 3: Saline Placebo
Started | 164 | 172 | 82
Completed | 159 | 170 | 81
Not Completed | 5 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Bupivacaine HCI | Treatment Group 3: Saline Placebo | Total
Number analyzed (Participants) | 164 | 172 | 82 | 418
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 149 | 161 | 77 | 387
  >=65 years | 15 | 11 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (13.29) | 49.4 (11.26) | 48.0 (14.59) | 48.9 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 3 | 23
  Male | 152 | 164 | 79 | 395
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 51 | 30 | 124
  Not Hispanic or Latino | 121 | 121 | 52 | 294
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 0 | 5
  Black or African American | 17 | 16 | 3 | 36
  White | 139 | 153 | 78 | 370
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 0 | 0 | 4
  United States | 160 | 172 | 82 | 414

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores With Activity (NRS-A) Through 72 Hours Postsurgery (AUC0-72), Compared With Saline Placebo.
Description: Pain intensity is assessed using an 11-point NRS (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable" (using windowed worst observation carried forward to adjust for opioid rescue medication use). The theoretical range of AUC0-72 is 0-720. The prescribed activity for NRS-A is sitting up from a resting position.
Time Frame: 72 hours
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 3: Saline Placebo
Number analyzed (Participants) | 164 | 82
pain intensity score*hr | 269.39 (173.719) | 350.82 (171.224)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 3: Saline Placebo; Test type: Superiority; p = 0.0004, ANOVA; Least Squares Mean Difference (LSMD) = -81.43, 95% CI 2-sided [-125.83 to -37.02], Standard Error of Mean 22.592

2. Secondary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores With Activity (NRS-A) Through 72 Hours Postsurgery (AUC0-72), Compared With Bupivacaine HCl.
Description: as for outcome 1
Time Frame: 72 hours
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Bupivacaine HCI
Number analyzed (Participants) | 164 | 172
pain intensity score*hr | 269.39 (173.719) | 341.88 (158.303)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 2: Bupivacaine HCI; Test type: Superiority; p < 0.0001, ANOVA; Least Squares Mean Difference (LSMD) = -72.49, 95% CI 2-sided [-108.32 to -36.65], Standard Error of Mean 18.23

3. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in Morphine Equivalents) for HTX 011 Compared With Saline Placebo.
Time Frame: 72 hours
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: IV milligram morphine equivalent (MME)
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 3: Saline Placebo
Number analyzed (Participants) | 164 | 82
IV milligram morphine equivalent (MME) | 10.85 (17.062) | 17.53 (18.908)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 3: Saline Placebo; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percetange of Subjects Who Are Opioid-free for HTX-011 Compared With Bupivacaine HCl.
Time Frame: 72 hours
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Bupivacaine HCI
Number analyzed (Participants) | 164 | 172
Participants | 84 | 69
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 2: Bupivacaine HCI; Test type: Superiority; p = 0.0486, Fisher Exact; Risk Difference (RD) = 0.111, 95% CI 2-sided [0.003 to 0.218]

5. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in Morphine Equivalents) for HTX 011 Compared With Bupivacaine HCl.
Time Frame: 72 hours
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: IV milligram morphine equivalent (MME)
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Bupivacaine HCI
Number analyzed (Participants) | 164 | 172
IV milligram morphine equivalent (MME) | 10.85 (17.062) | 14.51 (18.185)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 2: Bupivacaine HCI; Test type: Superiority; p = 0.024, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 28 days.
Description: For each Preferred Term (PT), subjects are included only once, even if they experienced multiple events in that PT.
Groups:
- Treatment Group 2: Bupivacaine HCI: Bupivacaine HCl without epinephrine, 75 mg by injection.
  173 = Safety Population because 1 subject was randomized to HTX-011, but received bupivacaine HCl.
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Bupivacaine HCI | Treatment Group 3: Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/173 | 0/82
Serious Adverse Events (participants affected / at risk) | 2/163 | 1/173 | 1/82
Other Adverse Events (participants affected / at risk) | 84/163 | 104/173 | 49/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: HTX-011 (N=163) | Treatment Group 2: Bupivacaine HCI (N=173) | Treatment Group 3: Saline Placebo (N=82)
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: HTX-011 (N=163) | Treatment Group 2: Bupivacaine HCI (N=173) | Treatment Group 3: Saline Placebo (N=82)
Nausea (Gastrointestinal disorders) | 30 | 37 | 28
Constipation (Gastrointestinal disorders) | 28 | 41 | 15
Dizziness (Nervous system disorders) | 24 | 42 | 13
Headache (Nervous system disorders) | 21 | 24 | 10
Bradycardia (Cardiac disorders) | 15 | 16 | 6
Dysgeusia (Nervous system disorders) | 15 | 21 | 3
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 13 | 1 | 1
Tremor (Nervous system disorders) | 7 | 12 | 8
Vomiting (Gastrointestinal disorders) | 7 | 12 | 4
Tinnitus (Ear and labyrinth disorders) | 3 | 6 | 5
Gamma-glutamyltransferase increase (Investigations) | 2 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03237481/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03237481/SAP_001.pdf